CLINICAL TRIAL: NCT06980831
Title: Developmental of Virtual Reality for Nursing Students: Electroconvulsive Therapy
Brief Title: Development of Virtual Reality for Nursing Students: Electroconvulsive Therapy
Acronym: Experimental
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mae Fah Luang University (Other)
Responsible Party: Principal Investigator, Chuntana Reangsing, School of Nursing, Mae Fah Luang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-24116-19
Record Dates: First submitted 2025-01-16; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Electroconvulsive Therapy; Knowledge, Attitudes, Practice
Keywords: knowledge; attitude; satisfaction; self-confidence; electroconvulsive therapy
MeSH Terms: conditions — Behavior; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): ECT group
  Interventions: Procedure: ECT group
- control group (No Intervention): waitlist control group

INTERVENTIONS:
Procedure: ECT group — VR-ECT group, nursing students will practice via virtual reality for taking care of patients with ECT.
  Arms: Experimental group

SUMMARY:
Project: "Development of virtual reality for nursing students: ECT"

For this project the researchers will adapte 'health belief model' as a core concept for developing knowledge, attitude and skills of nursing students to take care of psychiatric patients with ECT. For their practice, the participants will be taught to take care of patients with ECT into 3 phases: before, during, and after ECT.

The researchers believe that this VR technology will help Thai-nursing students better understand and know how to take care of patients with ECT.

This project will consist of two phase. phase I: developing VR- ECT technology for nursing students. we will pilot test VR-ECT in Nursing students by randomizing nursing students volunteers into two groups: an experimental group and waitlist control group (N = 140). Knowledge, attitude and satisfaction and self-confidence will be measured at baseline (day 1), week 8 after intervention complete

DETAILED DESCRIPTION:
Population: Thai nursing students who are between 18-24 years old who are studying in bachalor of Nursing, Thailand.

Sample:

Inclusion criteria: the researchers will include bachelor nursing students who 1) are between 18-24 year of age; 2) are proficient in Thai; 3) are never study in ECT class; and 4) volunteer.

Exclusion criteria: the researchers will exclude nursing students if they have 1) current presence of physical or mental condition such as learning disorders, and psychiatric disorders, all of which make full participation in all aspects of this study questionable; 2) already studies and had experienced with ECT nursing care.

Phase I: To develop the ECT virtual reality for nursing students

* 20 nursing students for VR-testing

Phase II: To evaluate the effects of VR-ECT for nursing students on knowledge, attitude, satisfaction and self-confidence among Thai-nursing students.

* Quantitative sample: 140 nursing students randomized to two groups to test the effectiveness and efficacy of the VR-ECT.
* Qualitative sample: 20 nursing students for in-depth interview and focus group to get the nursing students' experience and perception of VR-ECT.

ELIGIBILITY:
Inclusion Criteria:

* the researchers will include Thai-nursing students who 1) are between 18 and 24 years of age; 2) are proficient in Thai; 3) volunteer

Exclusion Criteria:

* the researchers will exclude Thai nursing students who 1) current presence of physical or mental conditions such as learning disorders and psychiatric disorders, all of which make full participation in all aspects of this study questionable; 2) had already studied in ECT or had experienced for taking care patients with ECT.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
VR-ECT knowledge (Thai version) | Day 1 -8 wk after intervention complete
  the researchers will adapt the knowledge for ECT nursing by Pruge and Vichai (2022) to measure the knowledge of nursing students for ECT nursing including the indication for ECT, Action and Side Effects, steps for ECT nursing, and adverse effect of ECT. The instrument including 18 items, each item has two options for yes (1 score) and no (o score).
VR-ECT attitude (Thai -version) | Day 1 - 8 week after intervention completed
  The researcher adapted questions developed by Pomporn Thongmuang (16). The purpose of this assessment was to measure nursing students' attitudes towards electrotherapy. It consists of 10 questions. The highest score indicates a positive attitude towards electroconvulsive therapy.
VR-ECT Satisfaction (Thai-version) | Day 1 - 8 week after intervention completed
  For the satisfaction on using VR-ECT technology (Satisfaction_VR-ECT) by Wanthana Pankamdee (17). The researcher will adapt this instrument based on the University students in Thailand context. The items including 40 items related with satisfaction of VR-ECT technology as Likert scale (1=dissatisfied to 5=very satisified). The high score indicates the high level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Chuntana Reangsing, PhD, RN, Principal Investigator — School of Nursing ,Mae Fah Luang University, Thailand

IPD SHARING:
Plan to Share IPD: Yes
No individual participant data will be shared. Results will be published by the investigators in academic journals. Sharing of generated study data will be carried out in several different ways. We plan to make our results available to researchers and potential collaborators interested in patients with ECT
Supporting Information: Study Protocol, SAP